CLINICAL TRIAL: NCT05187728
Title: Association Between the Occurrence of Adenomyosis and the Clinical Outcomes of Vaginal Repair ofCesareanSectionScar Defects:An Observational Study
Brief Title: Association Between the Adenomyosis and the Clinical Outcomes of Vaginal Repair of CesareanSectionScar Defects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-21-009
Record Dates: First submitted 2021-12-07; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Magnetic Resonance Imaging; Cesarean Section; Complications, Wound, Dehiscence
Keywords: Magnetic Resonance Imaging; cesarean scar defects; vaginal repair
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adenomyosis group: CSD with adenomyosis
  Interventions: Other: No Intervention
- non-adenomyosis group: CSD without adenomyosis
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No more intervention will be given.

SUMMARY:
To examine the correlation between the occurrence of adenomyosis and the outcome of vaginal repair of cesarean section scar defects (CSD), women with CSD will be enrolled in this retrospective observational cohort study. According to preoperative magnetic resonance imaging (MRI) findings, patients will be divided into two groups, the adenomyosis group and the non-adenomyosis group. They all will have vaginal excision and suture of CSD and will be required to undergo examinations at 3- and 6-months after surgery. Preoperative and postoperative clinical information will be collected.

DETAILED DESCRIPTION:
Women with CSD will be enrolled in this study. According to preoperative magnetic resonance imaging (MRI) findings, patients will be divided into two groups, the adenomyosis group and the non-adenomyosis group. They all underwent vaginal excision and suture of CSD and will be required to undergo examinations at 3- and 6-months after surgery. Preoperative and postoperative clinical information will be collected. Optimal healing was defined as a duration of menstruation of no more than 7 days and a TRM of no less than 5.30 mm after vaginal repair

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are non-pregnant patients who had one or more cesarean sections, patients who had intermenstrual spotting after the cesarean section or those in which the TRM was less than 3.0 mm at the preoperative stage, and patients who underwent MRI and TVS to evaluate the size of the defect and the TRM before surgery

Exclusion Criteria:

* Patients who had a history of chronic diseases (such as cerebro-cardiovascular diseases, malignancies and diabetes mellitus), endocrine disorders, menstrual irregularities before cesarean section, coagulation disorders, use of intrauterine devices, sub-mucous myoma, endometrial diseases, endometrial cysts, uterine fibroids, and adenomyosis after cesarean section

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Non-pregnant patients who had one or more cesarean sections, patients who had intermenstrual spotting after the cesarean section or those in which the TRM was less than 3.0 mm at the preoperative stage
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean duration of menstruation | on Days: 30
  Mean duration of menstruation
Mean duration of menstruation | on Days: 60
  Mean duration of menstruation
Mean duration of menstruation | on Days: 90
  Mean duration of menstruation
The thickness of the residual myometrium | on Days: 90
  The thickness of the residual myometrium

SECONDARY OUTCOMES:
reproductive information | 3 years
  reproductive information by questionnaire, including abortion, delivery, childbirth, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No